CLINICAL TRIAL: NCT00963820
Title: An Open-Label, Dose-Escalation, Phase 1 Study Evaluating the Safety and Tolerability of Weekly Dosing of the Oral Form of MLN9708, a Second-Generation Proteasome Inhibitor, in Adult Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Study Evaluating the Safety and Tolerability of Weekly Dosing of Oral IXAZOMIB in Adult Patients With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16004; U1111-1166-8401 (Other: WHO)
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed multiple myeloma; Refractory multiple myeloma; Drug therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- 0.24 mg/m^2 (Experimental): Ixazomib citrate, 0.24 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate
  Interventions: Drug: Ixazomib citrate
- 0.48 mg/m^2 (Experimental): Ixazomib citrate, 0.48 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- 0.80 mg/m^2 (Experimental): Ixazomib citrate, 0.80 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- 1.20 mg/m^2 (Experimental): Ixazomib citrate, 1.20 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period.
  Interventions: Drug: Ixazomib citrate
- 1.68 mg/m^2 (Experimental): Ixazomib citrate, 1.68 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- 2.23 mg/m^2 (Experimental): Ixazomib citrate, 2.23 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- 2.97 mg/m^2 (Experimental): Ixazomib citrate, 2.97 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- 3.95 mg/m^2 (Experimental): Ixazomib citrate, 3.95 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- Relapsed and Refractory (RR) (Experimental): Ixazomib citrate, 2.97 mg/m^2 established Maximum Tolerated Dose (MTD), capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the Relapsed and Refractory (RR) expansion cohort. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- VELCADE-Relapsed (VR) (Experimental): Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the VELCADE-relapsed (VR) expansion cohort. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- PI naïve (Experimental): Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in expansion cohort of participants who were proteasome inhibitor-naïve (PI naïve). All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate
- Carfilzomib (Experimental): Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the expansion cohort of participants who received their last dose of carfilzomib between 21 and 60 days prior to the first dose of ixazomib citrate. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
  Interventions: Drug: Ixazomib citrate

INTERVENTIONS:
Drug: Ixazomib citrate — Ixazomib citrate capsules
  Other Names: MLN9708

SUMMARY:
The primary objective of this study is to determine the safety profile, tolerability, and maximum tolerated dose of ixazomib citrate (MLN9708) when taken orally on a weekly dosing schedule by patients with relapsed and refractory multiple myeloma (RRMM). Secondary objectives include pharmacokinetics and response rates.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib citrate (MLN9708). Ixazomib citrate is being tested for people who have multiple myeloma who have relapsed after treatment or become unresponsive to treatment.

This study will determine the maximum tolerated dose (MTD) of ixazomib citrate using a dose escalation scheme. Once MTD is established, participants will be enrolled at MTD into one of the 4 expansion cohorts to characterize the safety, tolerability and efficacy of MLN9708. Blood samples for safety labs, hematology, serum chemistry and pharmacokinetic evaluations will be obtained at the timepoints specified. Disease response assessment is to be performed on the first day of every other cycle beginning with Cycle 3.

The study will enroll approximately 60 patients. All participants will receive treatment with ixazomib citrate. This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 60 days, and participants will make 12-16 visits to the clinic for study procedures.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following eligibility criteria to be enrolled in the study:

* Adult patients with multiple myeloma who have relapsed following at least 2 lines of therapy.
* Patients must have measurable disease.
* Appropriate functional status, including the recovery from the effects of prior antineoplastic therapy, and acceptable organ function as described in the protocol.
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse.
* Willing and able to give written informed consent.
* Suitable venous access for study-required blood sampling.

Exclusion Criteria:

* Peripheral neuropathy that is greater or equal to Grade 2.
* Major surgery or, serious infections, or infections that required systemic antibiotic therapy within 14 days before the first dose of study drug.
* Life-threatening illness unrelated to cancer.
* Diarrhea that is greater than Grade 1 as outlined in the protocol
* Systemic antineoplastic or radiation therapy within 14 days or cytotoxic agents, or treatment with any investigational products within 21 days before the first dose of study treatment.
* Treatment with any investigational proteasome inhibitor.
* Systemic treatment with prohibited medications that are outlined in the protocol within 14 days of study treatment.
* Ongoing therapy with corticosteroids greater than 10mg of prednisone or its equivalent per day.
* Central nervous system involvement.
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months.
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption of tolerance of IXAZOMIB including difficulty swallowing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - James R. Berenson, MD, Inc, West Hollywood, California
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Weill-Cornell Medical College, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Gupta N, Yang H, Hanley MJ, Zhang S, Liu R, Kumar S, Richardson PG, Skacel T, Venkatakrishnan K. Dose and Schedule Selection of the Oral Proteasome Inhibitor Ixazomib in Relapsed/Refractory Multiple Myeloma: Clinical and Model-Based Analyses. Target Oncol. 2017 Oct;12(5):643-654. doi: 10.1007/s11523-017-0524-3. PMID 28803351
- [Derived] Kumar SK, Bensinger WI, Zimmerman TM, Reeder CB, Berenson JR, Berg D, Hui AM, Gupta N, Di Bacco A, Yu J, Shou Y, Niesvizky R. Phase 1 study of weekly dosing with the investigational oral proteasome inhibitor ixazomib in relapsed/refractory multiple myeloma. Blood. 2014 Aug 14;124(7):1047-55. doi: 10.1182/blood-2014-01-548941. Epub 2014 Jun 5. PMID 24904120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty (60) participants took part in the study at 6 investigative sites in the United States from 31 October 2009 to database lock on 28 February 2013.
Pre-assignment Details: Participants with a diagnosis of multiple myeloma (relapsed and/or refractory) were enrolled in the dose escalation phase to determine maximum tolerated dose (MTD). Once the MTD was established, participants were enrolled at the MTD into 1 of the 4 expansion cohorts.
Groups:
- 1.20 mg/m^2: Ixazomib citrate, 1.20 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
- Relapsed and Refractory (RR): Ixazomib citrate, 2.97 mg/m^2 established Maximum Tolerated Dose (MTD), capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the Relapsed and Refractory (RR) expansion cohort that includes 2 participants from the dose escalation cohort 2.97 mg/m^2. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
- VELCADE-relapsed (VR): Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the VELCADE-relapsed (VR) expansion cohort that includes 1 participant from the dose escalation cohort 2.97 mg/m^2. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
Period: Dose Escalation Phase
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Started | 3 | 3 | 3 | 3 | 4 | 3 | 8 | 5 | 0 (Expansion cohorts were not part of Dose Escalation except as noted in comments.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 4 | 3 | 8 | 5 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Started | 0 (Dose escalation cohorts were not part of the Expansion Phase except as noted in comments.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 (Includes 2 participants from the dose escalation cohort 2.97 mg/m^2.) | 10 (Includes 1 participant from the dose escalation cohort 2.97 mg/m^2.) | 6 (Includes only participants who are proteasome inhibitor (PI)-naïve.) | 4 (Includes participants with last dose of carfilzomib 21 to 60 days before 1st ixazomib citrate dose.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (Participant was ongoing at the time of data cut off for analysis) | 1 (Participant was ongoing at the time of data cut off for analysis) | 1 (Participant was ongoing at the time of data cut off for analysis) | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9 | 5 | 4
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Overall Study: Safety Population
Arm/Group | Overall Study
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 56
  Missing | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 51
  Black or African American | 7
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 60
Height [Mean (Standard Deviation); unit: cm] — Height data was missing for 1 participant. Mean and standard deviation calculation is based on 59 participants.
  cm | 168.4 (9.34)
Weight [Mean (Standard Deviation); unit: kg] | 83.26 (18.106)
Body Surface Area at Baseline [Mean (Standard Deviation); unit: m^2] — Body Surface Area (BSA) was missing for 1 participant. Mean and standard deviation are based on 59 participants.
  m^2 | 1.96 (0.247)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events and Serious Adverse Events
Description: An Adverse Event is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
  A Serious Adverse Event (SAE) was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From the first dose through 30 days after last dose of ixazomib citrate or until the start of subsequent antineoplastic therapy (Up to 354 days)
Population: Safety Population included all randomized participants who received study drug.
Measure: Number; unit: participants
Groups:
- Relapsed and Refractory (RR): Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the Relapsed and Refractory (RR) expansion cohort that includes 2 participants from the dose escalation cohort 2.97 mg/m^2. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 8 | 5 | 11 | 10 | 6 | 4
participants | 3 | 3 | 2 | 3 | 4 | 3 | 8 | 5 | 11 | 10 | 6 | 4

2. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for MLN2238
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Days 1 and 15 of Cycle 1
Population: Participants from the Pharmacokinetic (PK) Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for calculation of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 5 | 4 | 7 | 8 | 5 | 3
ng/mL
  Cycle 1 Day 1 (n=1,1,2,1,3,2,5,4,5,8,5,3) | 3.010 (NA) — Can not be calculated for 1 participant. | 2.91 (NA) — Can not be calculated for 1 participant. | 5.75 (4.1083) | 15.10 (NA) — Can not be calculated for 1 participant. | 13.83 (9.7070) | 29.05 (11.1016) | 65.46 (29.3351) | 123.95 (79.2137) | 75.92 (30.3995) | 110.43 (62.7006) | 77.70 (37.9107) | 83.73 (87.8161)
  Cycle 1 Day 15 (n=3,1,3,2,2,1,2,1,5,5,4,3) | 3.64 (0.9616) | 4.64 (NA) — Can not be calculated for 1 participant. | 6.89 (5.1116) | 17.90 (8.6267) | 17.63 (12.6926) | 9.24 (NA) — Can not be calculated for 1 participant. | 100.55 (15.1339) | 134.00 (NA) — Can not be calculated for 1 participant. | 50.46 (22.6877) | 93.68 (52.7617) | 118.05 (54.2907) | 55.10 (41.5275)

3. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for MLN2238
Description: Tmax: Time to reach the maximum observed plasma concentration (Cmax), equal to time to Cmax. MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Days 1 and 15 of Cycle 1
Population: Participants from the PK Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for analysis of Tmax.
Measure: Median (Full Range); unit: hours
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 5 | 4 | 7 | 8 | 5 | 3
hours
  Cycle 1 Day 1 (n=1,1,2,1,3,2,5,4,5,8,5,3) | 1.50 [1.50 to 1.50] | 1.53 [1.53 to 1.53] | 1.52 [1.03 to 2.00] | 1.00 [1.00 to 1.00] | 1.52 [1.00 to 2.00] | 1.25 [1.00 to 1.50] | 1.00 [0.50 to 4.00] | 1.00 [0.53 to 1.50] | 2.00 [0.50 to 2.00] | 0.50 [0.50 to 2.00] | 1.00 [0.50 to 1.42] | 1.42 [1.00 to 1.53]
  Cycle 1 Day 15 (n=3,1,3,2,2,1,2,1,5,5,4,3) | 1.07 [1.00 to 2.00] | 0.50 [0.50 to 0.50] | 1.83 [1.00 to 2.00] | 1.00 [1.00 to 1.00] | 1.27 [1.00 to 1.53] | 8.00 [8.00 to 8.00] | 1.25 [0.50 to 2.00] | 1.03 [1.03 to 1.03] | 1.50 [1.00 to 4.03] | 1.00 [0.50 to 1.50] | 1.00 [0.50 to 1.50] | 1.03 [1.00 to 4.00]

4. Secondary Outcome: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for MLN2238
Description: AUC(0-168) is a measure of the area under the plasma concentration-time curve over the dosing interval (tau) (AUC[0-tau]), where tau is the length of the dosing interval - 168 hours in this study). MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Days 1 and 15 of Cycle 1
Population: Participants from the PK Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for calculation of AUC(0-168).
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 5 | 4 | 7 | 8 | 5 | 3
hr*ng/mL
  Cycle 1 Day 1 (n=0,0,0,0,2,1,3,4,3,5,4,3) | NA (NA) — No participants with evaluable data | NA (NA) — No participants with evaluable data | NA (NA) — No participants with evaluable data | NA (NA) — No participants with evaluable data | 258.00 (93.3381) | 598.00 (NA) — Can not be calculated for 1 participant. | 1269.67 (429.3837) | 1371.25 (725.1939) | 1793.33 (507.6744) | 854.20 (330.0745) | 750.25 (312.3890) | 813.67 (262.5649)
  Cycle 1 Day 15 (n=0,0,2,0,2,1,2,1,1,4,3,2) | NA (NA) — No participants with evaluable data | NA (NA) — No participants with evaluable data | 398.50 (45.9616) | NA (NA) — No participants with evaluable data | 663.00 (142.8356) | 868.00 (NA) — Can not be calculated for 1 participant. | 3100.00 (834.3860) | 1460.00 (NA) — Can not be calculated for 1 participant. | 3690.00 (NA) — Can not be calculated for 1 participant. | 1777.75 (958.4767) | 1549.00 (1027.6930) | 2075.00 (1025.3048)

5. Secondary Outcome: Accumulation Ratio: Day 15 AUC0-168 / Day 1 AUC0-168 for MLN2238
Description: MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Day 15 of Cycle 1
Population: Participants from the PK Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for calculation of accumulation ratio.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 3 | 2 | 2
unitless |  |  |  |  | 2.64 (0.3960) | 1.45 (NA) — Can not be calculated for 1 participant. | 2.25 (NA) — Can not be calculated for 1 participant. | 1.19 (NA) — Can not be calculated for 1 participant. | 2.25 (NA) — Can not be calculated for 1 participant. | 2.19 (0.8228) | 1.97 (0.5869) | 2.37 (0.2192)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz) for MLN2238
Description: Terminal elimination rate constant (λz) is the rate at which drugs are eliminated from the body and the values were used for calculation of T1/2. MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Day 15 of Cycle 1
Population: Participants from the PK Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for calculation of terminal elimination rate constant.
Measure: Mean (Standard Deviation); unit: 1/hour
Groups:
- 2.23 mg/m^2: Ixazomib citrate, 2.23 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day dose escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 3 | 4 | 2
1/hour |  |  | 0.000 (NA) — Can not be calculated for 1 participant. | 0.000 (0.0001) | 0.000 (0.0003) | 0.00 (NA) — Can not be calculated for 1 participant. | 0.00 (NA) — Can not be calculated for 1 participant. | 0.00 (NA) — Can not be calculated for 1 participant. | 0.00 (0.0019) | 0.00 (0.0014) | 0.01 (0.0019) | 0.01 (0.0003)

7. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for MLN2238
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma. MLN2238 is the complete hydrolysis product of the study drug ixazomib citrate (MLN9708).
Time Frame: Day 15 of Cycle 1
Population: Participants from the PK Analysis Population, all participants who had sufficient dosing data to calculate PK parameters, with data available for calculation of terminal phase elimination half-life.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 3 | 4 | 2
hour |  |  | 271.00 (NA) — Can not be calculated for 1 participant. | 190.50 (7.7782) | 189.00 (12.7279) | 175.00 (NA) — Can not be calculated for 1 participant. | 246.00 (NA) — Can not be calculated for 1 participant. | 165.00 (NA) — Can not be calculated for 1 participant. | 186.00 (84.8528) | 202.33 (63.0899) | 123.90 (39.4620) | 108.00 (4.2426)

8. Secondary Outcome: Emax: Maximum Inhibition
Description: A Whole Blood 20S Proteasome Inhibition Parameter. There were no subjects in the Pharmacodynamic (PD) Analysis Set for the 2.23 mg/m^2 cohort, so PD tables do not include that arm.
Time Frame: Days 1 and 15 of Cycle 1
Population: PD analysis Population included all participants who had sufficient dosing data to calculate PD parameters
Measure: Mean (Standard Deviation); unit: Percentage of inhibition
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 1 | 5 | 5 | 10 | 8 | 5 | 3
Percentage of inhibition | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported

9. Secondary Outcome: TEmax: Time of Occurrence of Emax
Time Frame: Days 1 and 15 of Cycle 1
Population: PD analysis population included all participants who had sufficient dosing data to calculate PD parameters
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 1 | 5 | 5 | 10 | 8 | 5 | 3
Hours | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported. | NA (NA) — Due to concerns about the third-party laboratory's performance of the 20S assay, accuracy of the data cannot be considered reliable, and therefore, is not being reported.

10. Secondary Outcome: Overall Response to Treatment With Ixazomib Citrate Based on Investigator's Evaluation Over Time
Description: Responses were based on International Myeloma Working Group Uniform Criteria. Complete Response (CR)=Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
  Partial Response (PR)= reduction in M-Protein ≥50% in serum and ≥90% in 24-hour urine. If M-protein unmeasurable, ≥50% decrease in difference of involved and uninvolved Free Light Chain (FLC). If M-protein and FLC unmeasurable, ≥50% reduction in plasma cells is required, if baseline bone marrow plasma cell ≥30%. And ≥50% reduction in the size of soft tissue plasmacytomas.
  Minimal Response (MR)= 25-49% reduction in serum paraprotein for 6 weeks. 50-89% reduction in 24 hour urinary light chain excretion for 6 weeks. For Non-secretory myeloma patients, 25-49 % reduction in plasma cells in bone marrow and trephine biopsy for a 6 weeks. 25-49% reduction in the size of soft tissue plasmacytomas. No increase in the size or number of lytic bone lesions.
Time Frame: Up to 354 days
Population: Response-Evaluable Population included all participants who had measurable disease at Baseline, had received at least 1 dose of study drug, and had at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 3 | 4 | 4 | 11 | 9 | 6 | 4
percentage of participants
  CR + PR | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 25 [0 to 81] | 25 [0 to 81] | 9 [0 to 41] | 22 [3 to 60] | 17 [0 to 64] | 25 [0 to 81]
  CR + PR + MR | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 25 [0 to 81] | 25 [0 to 81] | 18 [2 to 52] | 33 [7 to 70] | 17 [0 to 64] | 25 [0 to 81]

11. Primary Outcome: Neurotoxicity Grading
Description: Neurotoxicity is graded using participant responses to 11 functional questions on a 5-point scale, where 0=Not at all and 4=Very much, using the Functional Assessment of Cancer Therapy/Gynecology Oncology Group - Neurotoxicity Questionnaire, Version 4.0(14). Neurotoxicity subscale is a sum of 11 reversed item scores where each original score is transformed as (4 - score). The highest possible score is 44, and a higher score indicates more neurotoxicity.
Time Frame: Cycle 1 Day 1 and End of Study (Up to 354 days)
Population: Safety Population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.24 mg/m^2 | 0.48 mg/m^2 | 0.80 mg/m^2 | 1.20 mg/m^2 | 1.68 mg/m^2 | 2.23 mg/m^2 | 2.97 mg/m^2 | 3.95 mg/m^2 | Relapsed and Refractory (RR) | VELCADE-relapsed (VR) | PI naïve | Carfilzomib
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 8 | 5 | 11 | 10 | 6 | 4
score on a scale
  Cycle 1 Day 1 (n=2,3,3,3,4,3,7,4,9,8,6,4) | 36.00 (9.899) | 40.33 (1.155) | 42.00 (3.464) | 36.00 (7.937) | 39.50 (2.646) | 36.80 (4.530) | 33.14 (7.841) | 38.50 (4.203) | 38.44 (5.053) | 33.73 (6.935) | 38.00 (6.928) | 32.00 (8.367)
  End of Study (n=3,3,2,1,1,3,4,3,8,5,4,3) | 25.00 (3.606) | 40.67 (2.517) | 38.50 (3.536) | 35.00 (0.000) | 42.00 (0.000) | 36.00 (3.606) | 36.00 (7.528) | 33.33 (8.386) | 33.88 (9.219) | 27.24 (13.122) | 37.00 (5.944) | 27.33 (7.371)

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after last dose of ixazomib citrate or until the start of subsequent antineoplastic therapy (Up to 354 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Dose Escalation Cohorts: Ixazomib citrate, 0.24 to 3.95 mg/m^2, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the Dose Escalation period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
- Expansion Cohorts: Ixazomib citrate, 2.97 mg/m^2 established MTD, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the Expansion Period. All dose amounts are expressed as the dose of ixazomib, the biologically active moiety of ixazomib citrate.
Arm/Group | Dose Escalation Cohorts | Expansion Cohorts
Serious Adverse Events (participants affected / at risk) | 7/32 | 15/31
Other Adverse Events (participants affected / at risk) | 30/32 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohorts (N=32) | Expansion Cohorts (N=31)
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Stenosis or Obstruction of Ileus (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Hepatitis B (Infections and infestations) | 0 | 1
Abscess Neck (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohorts (N=32) | Expansion Cohorts (N=31)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Leukopenia (Blood and lymphatic system disorders) | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 6 | 10
Neutropenia (Blood and lymphatic system disorders) | 4 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 17
Lacrimation increased (Eye disorders) | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 4 | 6
Flatulence (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 2 | 4
Fatigue (General disorders) | 17 | 17
Influenza like illness (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 6
Cellulitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bicarbonate decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 6 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 6 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 7
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 5
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish clinical data after the earlier of publication by Sponsor or 12 months after early termination or database lock. Proposed publication copy should be provided to Sponsor at least 30 days prior to submission/disclosure. If requested, Sponsor's confidential information must be removed and publication delayed if Sponsor intends to file a related patent application.